CLINICAL TRIAL: NCT05798572
Title: Is Preoperative Sildosine Adminstration Faciltate Ureteral Diltation During Flexible Ureterorenoscopy?
Brief Title: Pre-Op Sildosine and Ureteral Dilation During F-URS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tamer Abd El-Wahab Diab, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ms: 7-12-2022
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: FURS; Ureteral Dilatation; Sildosine
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildosin group (Experimental): included 70 patients for whom flexible ureteroscopy (F-URS) was done with the daily preoperative intake of 8 mg silodosin for one week.
  Interventions: Drug: Sildosin group
- Placebo/control group (Experimental): included 70 patients for whom flexible ureteroscopy (F-URS) was done with daily preoperative intake of placebo tablets.
  Interventions: Procedure: Placebo/control group

INTERVENTIONS:
Drug: Sildosin group — Patients in this group had flexible ureteroscopy (F-URS) with preoperative daily uptake of 8 mg silodosin for one week.
  Arms: Sildosin group
Procedure: Placebo/control group — included 70 patients for whom flexible ureteroscopy (F-URS) was done with daily preoperative intake of placebo tablets.
  Arms: Placebo/control group

SUMMARY:
We proposed that silodosin administration preoperatively may facilitate ureteral access sheath (UAS) placement prior to flexible ureteroscopy (F-URS) and decrease the incidence of ureteric injury in some difficult cases.

DETAILED DESCRIPTION:
Urolithiasis is a common urological disorder in the world and has a significant effect on the global health system. The goal of treatment is to achieve the highest stone-free rate (SFR) with the least invasive. Per¬cutaneous nephrolithotomy and flexible ureterorenoscopy (F-URS) are the two main minimally invasive procedures for the treatment of upper urinary tract stones.

The challenging step in flexible ureterorenoscopy (F-URS) is ureteroscopic access sheath (UAS) placement, which facilitates fast and safe access to the ureter and collecting system; improves visibility; reduces the risk of infection by reducing intrarenal pressure. However, in some cases, the acute ureteric injury may occur during ureteroscopic access sheath (UAS) placement.

ELIGIBILITY:
Inclusion Criteria:

* Upper ureteric stone or stone kidney (with stone burden equal to or less than 20mm).
* 2. Non stented.
* Age (Above 18 years old).

Exclusion Criteria:

* Acute or chronic renal insufficiency.
* Uncorrected coagulopathy.
* Previous open (lumber or ureteric) surgery.
* Active urinary tract infection unless treated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Entrance to bladder time (ETBT) | Intraoperatively
  Entrance to bladder time (ETBT) will be recorded

SECONDARY OUTCOMES:
Entrance to ureteric orifice time (ETUOT) | Intraoperatively
  Entrance to ureteric orifice time (ETUOT) will be recorded
Application of access sheath time (AAST) | Intraoperatively
  Application of access sheath time (AAST) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study.